CLINICAL TRIAL: NCT03715621
Title: A Study of Prognostic Values of Next Generation Sequencing (NGS) in Acute Myeloid Leukemia Patients With Allo-HSCT
Brief Title: Prognostic Values of Next Generation Sequencing (NGS) in Acute Myeloid Leukemia Patients With Allo-HSCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Wu Depei, professor, The First Affiliated Hospital of Soochow University
Other Study IDs: AML-NGS-2018
Record Dates: First submitted 2018-09-27; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; next generation sequencing; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute myeloid leukemia (AML) is a genetically heterogeneous disease and allogeneic hematopoietic stem cell transplantation (allo-HSCT) is a curative treatment option for AML except for AML-M3. Relapse remains the major cause of treatment failure after allo-HSCT. Molecular residual disease has been shown to be a strong risk factor for relapse after HSCT. In this study, the investigators will detect mutations before/after allo-HSCT by using next-generation sequencing (NGS) technique to measure residual disease and evaluate the prognostic impact of molecular residual disease in a cohort of AML participants receiving allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or old;
* Clinical diagnosis of acute myeloid leukemia (AML);
* Availabe records of MICM and NGS results at diagnosis;
* Be going to receive allo-HSCT.

Exclusion Criteria:

* Active malignancy;
* Pregnant or breast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with the diagnosis of AML who is going to receive an allo-geneic HSCT within 30 days
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2020-10-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
1-year relapse rate after allo-HSCT | 1 year after allo-HSCT
  1-year relapse rate after allo-HSCT

SECONDARY OUTCOMES:
1-year recurrence-free survival (RFS) | 1 year after allo-HSCT
  1-year recurrence-free survival for AML participants
1-year overall survival (OS) | 1 year after allo-HSCT
  1-year overall survival (OS) for AML participants

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, doctor, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First affiliated Hospital of SooChow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dohner H, Weisdorf DJ, Bloomfield CD. Acute Myeloid Leukemia. N Engl J Med. 2015 Sep 17;373(12):1136-52. doi: 10.1056/NEJMra1406184. No abstract available. PMID 26376137
- [Background] Schmid C, Labopin M, Nagler A, Niederwieser D, Castagna L, Tabrizi R, Stadler M, Kuball J, Cornelissen J, Vorlicek J, Socie G, Falda M, Vindelov L, Ljungman P, Jackson G, Kroger N, Rank A, Polge E, Rocha V, Mohty M; Acute Leukaemia Working Party of the European Group for Blood and Marrow Transplantation (EBMT). Treatment, risk factors, and outcome of adults with relapsed AML after reduced intensity conditioning for allogeneic stem cell transplantation. Blood. 2012 Feb 9;119(6):1599-606. doi: 10.1182/blood-2011-08-375840. Epub 2011 Dec 13. PMID 22167752
- [Background] Corbacioglu A, Scholl C, Schlenk RF, Eiwen K, Du J, Bullinger L, Frohling S, Reimer P, Rummel M, Derigs HG, Nachbaur D, Krauter J, Ganser A, Dohner H, Dohner K. Prognostic impact of minimal residual disease in CBFB-MYH11-positive acute myeloid leukemia. J Clin Oncol. 2010 Aug 10;28(23):3724-9. doi: 10.1200/JCO.2010.28.6468. Epub 2010 Jul 12. PMID 20625124
- [Background] Yin JA, O'Brien MA, Hills RK, Daly SB, Wheatley K, Burnett AK. Minimal residual disease monitoring by quantitative RT-PCR in core binding factor AML allows risk stratification and predicts relapse: results of the United Kingdom MRC AML-15 trial. Blood. 2012 Oct 4;120(14):2826-35. doi: 10.1182/blood-2012-06-435669. Epub 2012 Aug 8. PMID 22875911
- [Background] Gorello P, Cazzaniga G, Alberti F, Dell'Oro MG, Gottardi E, Specchia G, Roti G, Rosati R, Martelli MF, Diverio D, Lo Coco F, Biondi A, Saglio G, Mecucci C, Falini B. Quantitative assessment of minimal residual disease in acute myeloid leukemia carrying nucleophosmin (NPM1) gene mutations. Leukemia. 2006 Jun;20(6):1103-8. doi: 10.1038/sj.leu.2404149. PMID 16541144
- [Background] Schnittger S, Kern W, Tschulik C, Weiss T, Dicker F, Falini B, Haferlach C, Haferlach T. Minimal residual disease levels assessed by NPM1 mutation-specific RQ-PCR provide important prognostic information in AML. Blood. 2009 Sep 10;114(11):2220-31. doi: 10.1182/blood-2009-03-213389. Epub 2009 Jul 8. PMID 19587375
- [Background] Kronke J, Schlenk RF, Jensen KO, Tschurtz F, Corbacioglu A, Gaidzik VI, Paschka P, Onken S, Eiwen K, Habdank M, Spath D, Lubbert M, Wattad M, Kindler T, Salih HR, Held G, Nachbaur D, von Lilienfeld-Toal M, Germing U, Haase D, Mergenthaler HG, Krauter J, Ganser A, Gohring G, Schlegelberger B, Dohner H, Dohner K. Monitoring of minimal residual disease in NPM1-mutated acute myeloid leukemia: a study from the German-Austrian acute myeloid leukemia study group. J Clin Oncol. 2011 Jul 1;29(19):2709-16. doi: 10.1200/JCO.2011.35.0371. Epub 2011 May 9. PMID 21555683
- [Background] Shayegi N, Kramer M, Bornhauser M, Schaich M, Schetelig J, Platzbecker U, Rollig C, Heiderich C, Landt O, Ehninger G, Thiede C; Study Alliance Leukemia (SAL). The level of residual disease based on mutant NPM1 is an independent prognostic factor for relapse and survival in AML. Blood. 2013 Jul 4;122(1):83-92. doi: 10.1182/blood-2012-10-461749. Epub 2013 May 8. PMID 23656730
- [Background] Cilloni D, Messa F, Arruga F, Defilippi I, Gottardi E, Fava M, Carturan S, Catalano R, Bracco E, Messa E, Nicoli P, Diverio D, Sanz MA, Martinelli G, Lo-Coco F, Saglio G. Early prediction of treatment outcome in acute myeloid leukemia by measurement of WT1 transcript levels in peripheral blood samples collected after chemotherapy. Haematologica. 2008 Jun;93(6):921-4. doi: 10.3324/haematol.12165. Epub 2008 Apr 28. PMID 18443273
- [Background] Cilloni D, Renneville A, Hermitte F, Hills RK, Daly S, Jovanovic JV, Gottardi E, Fava M, Schnittger S, Weiss T, Izzo B, Nomdedeu J, van der Heijden A, van der Reijden BA, Jansen JH, van der Velden VH, Ommen H, Preudhomme C, Saglio G, Grimwade D. Real-time quantitative polymerase chain reaction detection of minimal residual disease by standardized WT1 assay to enhance risk stratification in acute myeloid leukemia: a European LeukemiaNet study. J Clin Oncol. 2009 Nov 1;27(31):5195-201. doi: 10.1200/JCO.2009.22.4865. Epub 2009 Sep 14. PMID 19752335
- [Background] Najima Y, Ohashi K, Kawamura M, Onozuka Y, Yamaguchi T, Akiyama H, Sakamaki H. Molecular monitoring of BAALC expression in patients with CD34-positive acute leukemia. Int J Hematol. 2010 May;91(4):636-45. doi: 10.1007/s12185-010-0550-8. Epub 2010 Apr 8. PMID 20376583
- [Background] Ostergaard M, Olesen LH, Hasle H, Kjeldsen E, Hokland P. WT1 gene expression: an excellent tool for monitoring minimal residual disease in 70% of acute myeloid leukaemia patients - results from a single-centre study. Br J Haematol. 2004 Jun;125(5):590-600. doi: 10.1111/j.1365-2141.2004.04952.x. PMID 15147374
- [Background] Kern W, Voskova D, Schoch C, Hiddemann W, Schnittger S, Haferlach T. Determination of relapse risk based on assessment of minimal residual disease during complete remission by multiparameter flow cytometry in unselected patients with acute myeloid leukemia. Blood. 2004 Nov 15;104(10):3078-85. doi: 10.1182/blood-2004-03-1036. Epub 2004 Jul 29. PMID 15284114
- [Background] Al-Mawali A, Gillis D, Lewis I. The use of receiver operating characteristic analysis for detection of minimal residual disease using five-color multiparameter flow cytometry in acute myeloid leukemia identifies patients with high risk of relapse. Cytometry B Clin Cytom. 2009 Mar;76(2):91-101. doi: 10.1002/cyto.b.20444. PMID 18727068
- [Background] Buccisano F, Maurillo L, Gattei V, Del Poeta G, Del Principe MI, Cox MC, Panetta P, Consalvo MI, Mazzone C, Neri B, Ottaviani L, Fraboni D, Tamburini A, Lo-Coco F, Amadori S, Venditti A. The kinetics of reduction of minimal residual disease impacts on duration of response and survival of patients with acute myeloid leukemia. Leukemia. 2006 Oct;20(10):1783-9. doi: 10.1038/sj.leu.2404313. Epub 2006 Jul 13. PMID 16838027
- [Background] Grubovikj RM, Alavi A, Koppel A, Territo M, Schiller GJ. Minimal residual disease as a predictive factor for relapse after allogeneic hematopoietic stem cell transplant in adult patients with acute myeloid leukemia in first and second complete remission. Cancers (Basel). 2012 Jun 20;4(2):601-17. doi: 10.3390/cancers4020601. PMID 24213327
- [Background] Walter RB, Buckley SA, Pagel JM, Wood BL, Storer BE, Sandmaier BM, Fang M, Gyurkocza B, Delaney C, Radich JP, Estey EH, Appelbaum FR. Significance of minimal residual disease before myeloablative allogeneic hematopoietic cell transplantation for AML in first and second complete remission. Blood. 2013 Sep 5;122(10):1813-21. doi: 10.1182/blood-2013-06-506725. Epub 2013 Jul 11. PMID 23847197
- [Background] Walter RB, Gyurkocza B, Storer BE, Godwin CD, Pagel JM, Buckley SA, Sorror ML, Wood BL, Storb R, Appelbaum FR, Sandmaier BM. Comparison of minimal residual disease as outcome predictor for AML patients in first complete remission undergoing myeloablative or nonmyeloablative allogeneic hematopoietic cell transplantation. Leukemia. 2015 Jan;29(1):137-44. doi: 10.1038/leu.2014.173. Epub 2014 Jun 3. PMID 24888275
- [Background] Bastos-Oreiro M, Perez-Corral A, Martinez-Laperche C, Bento L, Pascual C, Kwon M, Balsalobre P, Munoz C, Buces E, Serrano D, Gayoso J, Buno I, Anguita J, Diez-Martin JL. Prognostic impact of minimal residual disease analysis by flow cytometry in patients with acute myeloid leukemia before and after allogeneic hemopoietic stem cell transplantation. Eur J Haematol. 2014 Sep;93(3):239-46. doi: 10.1111/ejh.12336. Epub 2014 Apr 29. PMID 24702162
- [Background] Anthias C, Dignan FL, Morilla R, Morilla A, Ethell ME, Potter MN, Shaw BE. Pre-transplant MRD predicts outcome following reduced-intensity and myeloablative allogeneic hemopoietic SCT in AML. Bone Marrow Transplant. 2014 May;49(5):679-83. doi: 10.1038/bmt.2014.9. Epub 2014 Feb 10. PMID 24510069
- [Background] Ustun C, Courville EL, DeFor T, Dolan M, Randall N, Yohe S, Bejanyan N, Warlick E, Brunstein C, Weisdorf DJ, Linden MA. Myeloablative, but not Reduced-Intensity, Conditioning Overcomes the Negative Effect of Flow-Cytometric Evidence of Leukemia in Acute Myeloid Leukemia. Biol Blood Marrow Transplant. 2016 Apr;22(4):669-675. doi: 10.1016/j.bbmt.2015.10.024. Epub 2015 Nov 10. PMID 26551635
- [Background] Araki D, Wood BL, Othus M, Radich JP, Halpern AB, Zhou Y, Mielcarek M, Estey EH, Appelbaum FR, Walter RB. Allogeneic Hematopoietic Cell Transplantation for Acute Myeloid Leukemia: Time to Move Toward a Minimal Residual Disease-Based Definition of Complete Remission? J Clin Oncol. 2016 Feb 1;34(4):329-36. doi: 10.1200/JCO.2015.63.3826. Epub 2015 Dec 14. PMID 26668349
- [Background] Klco JM, Miller CA, Griffith M, Petti A, Spencer DH, Ketkar-Kulkarni S, Wartman LD, Christopher M, Lamprecht TL, Helton NM, Duncavage EJ, Payton JE, Baty J, Heath SE, Griffith OL, Shen D, Hundal J, Chang GS, Fulton R, O'Laughlin M, Fronick C, Magrini V, Demeter RT, Larson DE, Kulkarni S, Ozenberger BA, Welch JS, Walter MJ, Graubert TA, Westervelt P, Radich JP, Link DC, Mardis ER, DiPersio JF, Wilson RK, Ley TJ. Association Between Mutation Clearance After Induction Therapy and Outcomes in Acute Myeloid Leukemia. JAMA. 2015 Aug 25;314(8):811-22. doi: 10.1001/jama.2015.9643. PMID 26305651
- [Background] Ten years of methods. Nat Methods. 2014 Oct;11(10):1000-1. doi: 10.1038/nmeth1014-1000. No abstract available. PMID 25264774
- [Background] Getta BM, Devlin SM, Levine RL, Arcila ME, Mohanty AS, Zehir A, Tallman MS, Giralt SA, Roshal M. Multicolor Flow Cytometry and Multigene Next-Generation Sequencing Are Complementary and Highly Predictive for Relapse in Acute Myeloid Leukemia after Allogeneic Transplantation. Biol Blood Marrow Transplant. 2017 Jul;23(7):1064-1071. doi: 10.1016/j.bbmt.2017.03.017. Epub 2017 Mar 15. PMID 28315400